CLINICAL TRIAL: NCT02170818
Title: Improving Faculty's Ability to Speak Up to Others in the Operating Room: A Simulation Based Randomized Controlled Trial of an Educational Intervention
Brief Title: Improving Faculty's Ability to Speak Up to Others in the Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Principal Investigator, Daniel Raemer, Ph.D., Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2008P001015
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Faculty, Medical
Keywords: Education; Curriculum; Anesthesiology; Operating Rooms
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Workshop on Speaking-Up (Experimental): Educational Workshop on Speaking-Up Before Simulated Case
  Interventions: Other: Educational Workshop on Speaking-Up
- Unrelated Education (Sham Comparator): Unrelated Education (CPR) before simulated case (Educational Workshop on Speaking-up after case and debriefing)
  Interventions: Other: Unrelated Education (CPR)

INTERVENTIONS:
Other: Educational Workshop on Speaking-Up — Educational workshop including lecture, discussion, role-play Concepts include: 2-challenge rule, pairing advocacy and inquiry
  Arms: Educational Workshop on Speaking-Up
Other: Unrelated Education (CPR) — Unrelated Education (CPR workshop) including: lecture, discussion Topics covered: Cardiac Life Support algorithms, CPR, Medications
  Arms: Unrelated Education

SUMMARY:
Importance Team members speaking-up by raising concerns about inappropriate or unsafe actions of others within the team can have direct, immediate, and preventive effect on adverse outcomes. However, little is known about the hurdles and enablers of this behavior in healthcare, especially within the operating room setting.

Objective

1. Determine if an educational workshop would improve speaking-up behaviors of practicing anesthesiologists when presented with realistically-simulated clinical situations. 2.Describe speaking-up behaviors addressed to a surgeon, a nurse, and a colleague. 3. Identify the self-reported hurdles and enablers for speaking-up in those situations encountered.

Design Randomized controlled experiment of an educational workshop intervention on communication behaviors in a simulated case. Qualitative analysis of debriefing conversations following the simulated case.

Setting Established academic simulation center

Participants Seventy-one practicing anesthesiologists from four academic medical centers and one community hospital

Intervention Fifty minute educational workshop on speaking-up that included rationale, conversational techniques, a rubric for speaking-up, and role-play.

DETAILED DESCRIPTION:
Main Outcomes and Measures

1. Observed communication in a simulated case that included a surgeon falling asleep during surgery, inappropriate activation of a speakerphone by a nurse, and an incorrect treatment order by a colleague in response to a venous air embolism. 2. Transcribed conversation during a structured debriefing, analyzed for hurdles and enablers.

ELIGIBILITY:
Inclusion Criteria:

* Attending Anesthesiologist

Exclusion Criteria:

* Prior exposure to test case

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2008-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Speaking-Up Behavior | Immediate
  Subjects were assessed by trained raters as to whether they spoke-up when safety related errors were made during a realistic simulation case.

SECONDARY OUTCOMES:
Speaking-up Behaviors | Immediate
  Anesthesiologist subject's behavior in speaking-up to a surgeon, nurse, and colleague during a realistic simulation case were assessed descriptively.
Self-reported hurdles and enablers of speaking-up | 1 hour
  A qualitative analysis of stated hurdles or enablers for speaking-up or not was conducted from video recordings of a post-case structured debriefing.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Raemer, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States